CLINICAL TRIAL: NCT03023059
Title: Proof of Concept and Dose Ranging Study of Carbidopa-levodopa in Neovascular AMD
Brief Title: Dose Ranging Study of Carbidopa-levodopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Snyder, Robert W., M.D., Ph.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0002
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Age-related Macular Degeneration
Keywords: L-DOPA; GPR143; PEDF; VEGF
MeSH Terms: conditions — Macular Degeneration | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Escalating dose of carbidopa-levodopa (Experimental): The intervention is that patients will receive open label, commercially available Carbidopa-Levodopa 25 Mg-100 Mg oral tablet, once daily hs for one month, followed by one tablet dosed three times daily, in the morning, with supper and hs for one month, followed by two tablets dosed three times daily, in the morning, with supper and hs for one month (100-600 mg of levodopa daily). This is the equivalent of very low to moderate doses of carbidopa-levodopa in patients with Parkinson's disease (daily dose of levodopa 200-800 mg).
  Interventions: Drug: Carbidopa-Levodopa, 25 Mg-100 Mg Oral Tablet

INTERVENTIONS:
Drug: Carbidopa-Levodopa, 25 Mg-100 Mg Oral Tablet — See Arm description
  Other Names: Sinemet

SUMMARY:
From 3 large patient databases, patients diagnosed with AMD who have never taken levodopa(L-DOPA) containing medications have a mean age of diagnosis at 71 years. Patients who have been treated with L-DOPA containing medications have a mean age of diagnosis of AMD at 79 years.

L-DOPA binds to GPR143 in the retinal pigment epithelium, and releases PEDF, which protects the retina and downregulates VEGF, which is the cause of neovascularization.

The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with Neovascular AMD, and measure the effects on visual acuity and retinal abnormalities due to "wet" (neovascular) AMD.

The Investigators will evaluate the safety and tolerability of carbidopa-levodopa in patients with Neovascular AMD who are already on treatment with anti-VEGF intraocular injections, and measure the effects on visual acuity, retinal abnormalities due to "wet" AMD, and document the number of anti-VEGF injections required during the study.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is the most common cause of blindness, in individuals over the age of 50, in the developed world. AMD becomes more common as people age and is more common in lightly pigmented individuals. AMD appears more common in patients with Parkinson's Disease than in those without. The AREDS nutritional supplements are effective in slowing the progress of intermediate AMD(5). Most AMD is "dry AMD", which progresses relatively slowly and may impair vision, but usually does not lead to legal blindness. There are two forms of AMD, "wet AMD" and geographic atrophy (GA), that can cause more profound vision loss. In aggregate, they occur in about 25% of patients with AMD. Wet AMD is due to new growth of abnormal blood vessels under the retina. The new blood vessels are believed to be due to an excessive release of vascular endothelial growth factor (VEGF) by the retinal pigment epithelium(RPE) cells. Wet AMD is now effectively treated with intraocular injections of VEGF inhibitors. Geographic Atrophy, the other form of advanced AMD, represents focal death of the RPE cells and overlying neurosensory retina. There is no current treatment for GA. It is suspected that GA is due in part to a localized inflammatory response, damage to RPE cells, and loss of RPE cell function. It may also be speculated that stimulation of RPE cells to release a potent neurotrophic factor, pigment epithelium derived factor (PEDF) may slow the progression of GA.

In 2008, Dr. Brian McKay identified a receptor, G protein coupled receptor #143(GPR143), on the surface of RPE cells and discovered that L-DOPA was the natural ligand or stimulator of GPR143. Dr. McKay showed that treatment of RPE cells with exogenous L-DOPA resulted in the release of additional PEDF. In subsequent work, Dr. McKay's group also showed that L-DOPA stimulation of PEDF in RPE cells was also associated with a decrease in VEGF. Thus, Dr McKay hypothesized that exogenous L-DOPA may prevent the onset of AMD or progression to wet AMD.

In 2015, Dr McKay and his associates published a paper that showed that patients, who had been treated with L-DOPA, had a delay in the onset of AMD by 8 years, compared to patients who had not been treated with L-DOPA. In addition, those who had AMD and went on to develop wet AMD did so 5 years later than those with no history of L-DOPA treatment. L-DOPA is an intermediate in the pigmentation pathway. Dr. McKay and his associates suggested that the reason darkly pigmented races do not get AMD nearly as frequently as lighter-pigmented races is that they produce more pigment, and thus more L-DOPA to stimulate GPR143 on RPE cells. According to this hypothesis, the stimulated RPE cells release PEDF and decrease VEGF, which together are responsible for the protective effect.

Pharmacology of L-DOPA and carbidopa:

L-DOPA is formed by 3-hydroxylation of tyrosine by tyrosine-3-monooxygenase (tyrosinase).(18) The primary metabolic pathway of L-DOPA is decarboxylation by amino acid decarboxylase to dopamine, which is responsible for most, but not all, of its pharmacologic effects and toxicity. When carbidopa is administered with L-DOPA, systemic levels of L-DOPA double, and central nervous system (CNS) L-DOPA increases from about 1% of the administered dose to about 4%. Levodopa freely passes from the systemic circulation into the retina and brain, but dopamine and carbidopa do not. Adverse events are markedly decreased when carbidopa is administered with L-DOPA, because systemic levels of the toxic metabolite of L-DOPA, dopamine, are markedly reduced. In most patients, 25 mg of carbidopa is sufficient to control side effects of 100 mg of L-DOPA, primarily nausea, by 90%.

L-DOPA is the natural ligand for GPR143 in the RPE cells. The Investigators' intent is to increase the L-DOPA available to RPE surface receptors (GPR 143) while minimizing peripheral toxicity. This concept is unique, because all other uses of L-DOPA rely on CNS conversion of L-DOPA to dopamine, in order to produce the desired effect.

Pathogenesis of Neovascular AMD.

Excess VEGF is the mediator of retinal neovascularization and other retinal pathological changes in "wet" AMD. Intraocular injections of anti-VEGF antibodies is the standard of care in "Wet" AMD. Several publications, including Lim et al, show that with careful monitoring of the visual acuity and retinas of patients with wet AMD, if there is no progression, there are no long-term adverse consequences of delaying initiation of anti-VEGF therapy for up to 4 weeks. The patients will all have had anti-VEGF therapy initiated. The patients will be monitored at monthly intervals, for up to 3 months, for indications for administration of anti-VEGF injections.

Since there are no established animal models for AMD, and L-DOPA has a good safety profile in healthy volunteers and patients with Parkinson's disease, the Investigators propose a prospective experiment to determine the safety and tolerability of L-DOPA, in a population of patients with AMD. The participants will be made aware of potential side effects of L-DOPA, which are listed in the Informed Consent, during the consent process. Adverse events will be elicited by questioning the participants at each visit. The participants will also be advised to call the site if they have any medical problems between visits.

The Investigators will also use this study to examine whether L-DOPA has a positive effect on visual acuity and pathologic retinal changes of "wet" AMD. The parameters to be evaluated are best corrected ETDRS visual acuity, macular thickness by spectral domain optical coherence tomography (SD OCT), new blood (hemorrhage) by direct retinal examination, or subjective decrease in vision.

Treatments:

Patients will receive open-label, commercially available carbidopa-levodopa 25-100 mg, one tablet once daily hs for one month, followed by one tablet dosed TID (three times daily), in the morning, with supper and hs for one month, followed by two tablets dosed three times daily, in the morning, with supper and hs for one month (100-600 mg of levodopa daily). This is the equivalent of very low to moderate doses of carbidopa-levodopa in patients with Parkinson's disease (daily dose of levodopa 200-800 mg). Patients entering this study after completing Study 001 will receive one month of the dose that he or she received in Study 001, and one month each of any doses higher than the dose that he or she received in Study 001.

Examples:

1. If the patient received carbidopa-levodopa 25-100 mg once daily in Study 001, he or she will receive one month of treatment with each of the 3 daily doses of carbidopa-levodopa.
2. If the patient received carbidopa-levodopa 25-100 mg TID in Study 001, he or she will receive one month of carbidopa-levodopa 25-100 mg TID, followed by one month of carbidopa-levodopa 25-100 mg, 2 tablets TID.

Each patient will receive an injection of anti-VEGF medication on the day carbidopa-levodopa dosing begins in this study. Each patient will be evaluated at monthly (25-35 day) intervals and injected or not, based upon the criteria listed below, which are based on clinical practice standard of care.

Criteria for anti-VEGF injections

All patients will have had at least one anti-VEGF intraocular injection prior to entering the study. Additional injections will be based on: monthly evaluation of ETDRS (Early Treatment Diabetic Retinopathy Study), visual acuity (decrease of 5 letters from previous visit); increased macular thickness (compared to normal and previous visit as measured by SD OCT; new blood (hemorrhage) on direct retinal examination; or subjective decrease in vision. If any of these criteria are met, or if, in the opinion of the Ophthalmologist, the patient requires anti-VEGF therapy, the patient will have an anti-VEGF intraocular injection. If none of these criteria are met at visits 2, 3, or 4, with patient agreement, anti-VEGF injection will not be done, and the patient will be reevaluated in 1 month. The study will end at Visit 5, and patients will begin standard of care treatment with anti-VEGF injections. Patients who have completed Study 0001, Short-term effects of carbidopa-levodopa in Neovascular AMD, will be eligible to enroll in the current study, Study 0002, Proof of Concept and Dose Ranging Study of carbidopa-levodopa in Neovascular AMD.

Number of subjects: 52 completed Duration: up to 112 days of treatment. Primary Endpoint: A statistically significant improvement (5 letters) by carbidopa-levodopa treatment in ETDRS visual acuity.

Measurements and Activities:

1. Informed Consent at Baseline;
2. Ophthalmic history and comprehensive eye examination; including visual acuity, wearing any prescription lenses, using an EDTRS chart, in both eyes prior to randomization, and ophthalmoscopic examination, and SD OCT;
3. Repeat assessment of visual acuity using an EDTRS chart, ophthalmoscopic examination, and SD OCT at monthly visits;
4. Demographics at Baseline;
5. Medical History, Vital Signs and Physical Examination at Baseline;
6. ECG, CBC (complete blood count), Chem 20 and HbA1C at Baseline;
7. Dispense study medication at visits 2, 3 and 4;
8. Pill count at visits 3, 4 and 5;
9. Non-directed assessment of adverse events at each visit, including classification as to severity, seriousness and body system.
10. Concomitant medications at each visit.
11. If a patient had the baseline evaluation in Study 001, that will be used as the baseline evaluation for this study.

Statistics: Descriptive statistics will be generated for, at a minimum, ETDRS visual acuity, central retinal thickness, amount of intraretinal and subretinal fluid and presence of hemorrhage. Within patient trajectories for these outcomes will be plotted, incorporating information on dose and duration. Due to the small sample size, model-based analyses will be considered only to be exploratory. Analysis of Variance may be conducted to relate logarithm of dose and duration of treatment to the outcomes listed above.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of AMD with choroidal neovascularization (CNV) in one eye;
2. a. Not previously treated with anti-VEGF injections; or

   b. On anti-VEGF injections for at least 3 months, and meets criteria for a repeat injection; or

   c. Patients, who have completed Study 001, may enter this trial at the point of initiation of the month of treatment with the dose of carbidopa-levodopa, that they received in Study 001;
3. Normal or dry AMD of any grade in the second eye;
4. Willingness to maintain AREDS vitamin supplements throughout the study, or remain off these supplements for the duration of the study, if not taking them prior to the study;
5. Informed Consent at Baseline.

Exclusion Criteria:

1. Any current use of L-DOPA containing medication or dopamine agonist medication, or any planned use of any of these agents, except for study medication, during the study;
2. Concurrent use of monoamine oxidase (MAO) inhibitors;
3. Any eye condition, disease, or history of trauma in either eye, which can impair vision, except cataract or cataract surgery;
4. Best Corrected Visual Acuity (BCVA) worse than 20/60 in the better eye;
5. Wet AMD in the second eye;
6. Neurologic conditions which can impair vision;
7. Parkinson's Disease;
8. Significant orthostatic hypotension, defined as a drop in systolic blood pressure, immediately upon changing from the supine to standing position, of >19 mmHg, or a symptomatic drop in systolic blood pressure, immediately upon changing from the supine to standing position;
9. Significant ECG abnormalities, as judged by the Investigator;
10. Estimated glomerular filtration rate (eGFR) <20 ml/min;
11. Liver enzymes >3 X the upper limit of normal;
12. HbA1C >9.0;
13. Any other significant lab abnormalities, as judged by the Investigator;
14. Women of childbearing potential;
15. Known retinal hemorrhage;
16. Subjects who are not fluent in English. -

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Snyder, MD, PhD, Principal Investigator — Robert W Snyder, MD, PhD, PC; Timothy C Fagan, MD, Study Director — Robert W Snyder, MD, PhD, PC
Locations (1):
- Robert W Snyder, MD, PhD, PC, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Background] Jager RD, Mieler WF, Miller JW. Age-related macular degeneration. N Engl J Med. 2008 Jun 12;358(24):2606-17. doi: 10.1056/NEJMra0801537. No abstract available. PMID 18550876
- [Background] Bressler SB, Munoz B, Solomon SD, West SK; Salisbury Eye Evaluation (SEE) Study Team. Racial differences in the prevalence of age-related macular degeneration: the Salisbury Eye Evaluation (SEE) Project. Arch Ophthalmol. 2008 Feb;126(2):241-5. doi: 10.1001/archophthalmol.2007.53. PMID 18268216
- [Background] Ferrara N. Vascular endothelial growth factor and age-related macular degeneration: from basic science to therapy. Nat Med. 2010 Oct;16(10):1107-11. doi: 10.1038/nm1010-1107. No abstract available. PMID 20930754
- [Background] Lopez VM, Decatur CL, Stamer WD, Lynch RM, McKay BS. L-DOPA is an endogenous ligand for OA1. PLoS Biol. 2008 Sep 30;6(9):e236. doi: 10.1371/journal.pbio.0060236. PMID 18828673
- [Background] Falk T, Congrove NR, Zhang S, McCourt AD, Sherman SJ, McKay BS. PEDF and VEGF-A output from human retinal pigment epithelial cells grown on novel microcarriers. J Biomed Biotechnol. 2012;2012:278932. doi: 10.1155/2012/278932. Epub 2012 Apr 2. PMID 22547925
- [Background] Brilliant MH, Vaziri K, Connor TB Jr, Schwartz SG, Carroll JJ, McCarty CA, Schrodi SJ, Hebbring SJ, Kishor KS, Flynn HW Jr, Moshfeghi AA, Moshfeghi DM, Fini ME, McKay BS. Mining Retrospective Data for Virtual Prospective Drug Repurposing: L-DOPA and Age-related Macular Degeneration. Am J Med. 2016 Mar;129(3):292-8. doi: 10.1016/j.amjmed.2015.10.015. Epub 2015 Oct 30. PMID 26524704
- [Background] Westfall TC, Westfall DP. Neurotransmission: The Autonomic and Somatic Nervous Systems. Pharmacological Basis of Therapeutics, 12th Edition, 171-218, McGraw-Hill, 2011.
- [Background] Standaert DG, Roberson ED. Treatment of Central Nervous System Degenerative Disorders. Pharmacological Basis of Therapeutics, 12th Edition, 609-628, McGraw-Hill, 2011
- [Background] Lim JH, Wickremasinghe SS, Xie J, Chauhan DS, Baird PN, Robman LD, Hageman G, Guymer RH. Delay to treatment and visual outcomes in patients treated with anti-vascular endothelial growth factor for age-related macular degeneration. Am J Ophthalmol. 2012 Apr;153(4):678-86, 686.e1-2. doi: 10.1016/j.ajo.2011.09.013. Epub 2012 Jan 14. PMID 22245460

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Escalating Dose of Carbidopa-levodopa
Started | 35
Completed | 30
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: This population includes participants who completed NCT03022318 (naive to anti-vascular endothelial growth factor injections at the time of enrollment) and patients who did not complete NCT03022318 but had been exposed to anti-VEGF injections before study initiation.
Groups:
- Escalating Dose of Carbidopa-levodopa: The intervention is that patients will receive open label, commercially available Carbidopa-Levodopa 25 Mg-100 Mg oral tablet, once daily at bedtime for one month, followed by one tablet dosed three times daily, in the morning, with supper and at bedtime for one month, followed by two tablets dosed three times daily, in the morning, with supper and bedtime for one month (100-600 mg of levodopa daily). This is the equivalent of very low to moderate doses of carbidopa-levodopa in patients with Parkinson's disease (daily dose of levodopa 200-800 mg).
  Carbidopa-Levodopa, 25 Mg-100 Mg Oral Tablet: See Arm description
Arm/Group | Escalating Dose of Carbidopa-levodopa
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 28
Age, Continuous [Mean (Full Range); unit: years] | 75.1 [58.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Patients naive to anti-VEGF injections at start of study [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity by Early Treatment Diabetic Retinopathy Study Chart Visual Scale Testing
Description: This outcome is a measure of letters correctly identified using an Early Treatment Diabetic Retinopathy Study chart. The higher the number of letters identified, the better the participant's visual acuity.
Time Frame: From the start of the study to the end (up to 120 days).
Population: This population includes participants who completed NCT03022318 (naive to anti-VEGF injections at the time of enrollment) and patients who did not complete NCT03022318 but had been exposed to anti-VEGF injections before study initiation.
Measure: Mean (Standard Error); unit: Change in letters (BCVA)
Arm/Group | Escalating Dose of Carbidopa-levodopa
Number analyzed (Participants) | 30
Change in letters (BCVA) | 4.5 (1.4)

2. Secondary Outcome: Change in Central Retinal (Macular) Thickness
Description: Central retinal thickness (in microns) is measured by spectral domain-optical coherence tomography. An increase in retinal thickness is associated with disease progression. A negative value represents a decrease in retinal thickness and therefore a positive clinical outcome measure.
Time Frame: From the start of the study to the end (up to 120 days).
Population: as for outcome 1
Measure: Mean (Standard Error); unit: microns
Arm/Group | Escalating Dose of Carbidopa-levodopa
Number analyzed (Participants) | 30
microns | -15.0 (9.8)

3. Secondary Outcome: Percent Change in Retinal Fluid From Baseline
Description: Retinal fluid changes on direct retinal examination on spectral domain - optical coherence tomography. Changes in retinal fluid were compared to baseline values. A negative percentage point represents a decrease in retinal fluid and therefore a positive clinical outcome.
Time Frame: From the start of the study to the commonly used timeframe of 6 months (~192 days), given that fluid was assessed at 6 months from baseline as commonly evaluated in studies involving AMD.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Escalating Dose of Carbidopa-levodopa
Number analyzed (Participants) | 30
percent change | 11.2 (30.6)

4. Secondary Outcome: Treatment Emergent Adverse Events
Description: Vital signs, eye examinations and nondirected subjective adverse events (gastrointestinal distress, muscle spasms, headache, nightmares)
Time Frame: From the start of the study to the commonly used timeframe of 6 months (~192 days), given that fluid was assessed at 6 months, we opted to include the evaluation of adverse events within the six months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Escalating Dose of Carbidopa-levodopa
Number analyzed (Participants) | 30
Participants | 9

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Escalating Dose of Carbidopa-levodopa
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 9/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Escalating Dose of Carbidopa-levodopa (N=30)
Mild malaise/nausea (General disorders) | 5
Mild-to-moderate back muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain and gas (Gastrointestinal disorders) | 2
Nightmares and mild headache (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
The major limitations of our study include the small sample size and limited patient racial diversity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-06-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT03023059/Prot_000.pdf